CLINICAL TRIAL: NCT05588362
Title: Access to EyeGlasses for School-aged Children
Acronym: ATEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Fitz Frames, Inc. (Unknown)
Responsible Party: Principal Investigator, Emily Wiecek, Optometrist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-P00040587
Record Dates: First submitted 2022-10-03; First posted 2022-10-20 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Myopia; Amblyopia; Hyperopia; Refractive Errors
MeSH Terms: conditions — Myopia; Amblyopia; Hyperopia; Refractive Errors

STUDY DESIGN:
Intervention Model Description: Prospective randomized control study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators responsible for administering questionnaires and collecting visual outcomes will be masked to the treatment group of the participant. Both the research assistant and participant will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitz Frames 3-D Printed Glasses (Experimental): The intervention group will order glasses directly in the office following their exam and consent using an iPad with the help of the research assistant. The iPad will be e-connected to a 3D printed glasses manufacturer (Fitz Frames) through their application, allowing the child (with assistance from the doctor or research assistant) to take various measurements in real time. Sixteen different measurements will be taken including interpupillary distance, face length, face width, and temple measures. The child will be able to choose frame style and order it directly from the manufacturer immediately following the exam. Glasses will be shipped directly to the patient's home (shipping address will be input to the app by the family).
  Interventions: Other: Fitz Frames 3-D Printed Glasses
- Traditional Glasses Procurement Group (No Intervention): (1) The control group will receive standard of care in which a prescription for glasses will be dispensed as a paper copy prescribed by the examiner before randomization. The research assistant will use a script (attached) that instructs families how to procure glasses traditionally through Masshealth. The participant/family will be instructed to bring the paper prescription to an optical shop that carries MassHealth frames. A printout of local optical shops that carry MassHealth frames will be provided to the patient.

INTERVENTIONS:
Other: Fitz Frames 3-D Printed Glasses — The intervention group will order glasses directly in the office following their exam and consent using an iPad with the help of the research assistant. The iPad will be e-connected to a 3D printed glasses manufacturer (Fitz Frames) through their application, allowing the child (with assistance from the doctor or research assistant) to take various measurements in real time. Sixteen different measurements will be taken including interpupillary distance, face length, face width, and temple measures. The child will be able to choose frame style and order it directly from the manufacturer immediately following the exam. Glasses will be shipped directly to the patient's home (shipping address will be input to the app by the family).
  Arms: Fitz Frames 3-D Printed Glasses

SUMMARY:
Uncorrected refractive error is a leading cause of visual impairment in children and can impact vision, quality of life, and academic performance. Despite Boston Children's Hospital serving patients from a wide range of socioeconomic backgrounds, there are health disparities in access to eyeglasses as a consequence of patients' health insurance. The investigators will examine whether the use of an in-clinic app for 3-D printed glasses reduces disparities in access to eyeglasses for our patients on Medicaid. The intervention will address social determinants of health and improve pediatric health outcomes namely, how and when children having publicly funded health insurance receive eyeglasses. The short-term objectives are (1) to compare the time to receive glasses between publicly funded MassHealth eyeglasses and an in-clinic order of 3D printed glasses (2) to evaluate compliance with glasses wear in these two groups, and (3) to evaluate visual function and quality-of-life outcomes in these two groups. This prospective randomized control study will evaluate barriers to accessing eyeglasses in school-aged children. The investigators will recruit children enrolled in MassHealth and randomize them into two cohorts: (1) the control group will receive MassHealth glasses as per standard of care, through an optical shop of their choosing, or (2) the intervention group will use an app for immediately ordering glasses (paid for by the study) in clinic following their appointment. The investigators will evaluate the time needed to receive eyeglasses, compliance with glasses wear, quality of life, and visual outcomes between the cohorts at one-, three-, and six-month intervals. Through this project, the investigators will not only evaluate, quantify, and bring awareness to disparities in our patient population, but will also look toward finding a solution through the use of a novel application that addresses many of the barriers faced by patients insured through Medicaid.

ELIGIBILITY:
Inclusion Criteria:

* Masshealth insurance
* first-time glasses wearers
* receive a diagnosis of refractive amblyopia, myopia, hyperopia and/or astigmatism requiring spectacle correction for optimal vision at distance and near.
* Glasses must be recommended for full time wear by the attending optometrist or ophthalmologist

Exclusion Criteria:

* strabismus
* developmental or learning delay
* other ocular pathology

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Compliance | Six months
  Glasses compliance will be assessed with self-reported calendar
Quality of Life Questionnaire | Baseline, will be collected at enrollment visit
  Quality of life measures using the PedEyeQ
Distance visual acuity | Baseline, will be collected at enrollment visit
  Linear Snellen optotypes (age >6) or HOTV matching with crowding bars (age <6)
Distance visual acuity | 0-3 Months, will be collected at 3 month visit
  Linear Snellen optotypes (age >6) or HOTV matching with crowding bars (age <6)
Distance visual acuity | 3-6 Months, will be collected at 6 month visit
  Linear Snellen optotypes (age >6) or HOTV matching with crowding bars (age <6)
Stereoacuity | Baseline, will be collected at enrollment visit
  Stereo Fly test
Stereoacuity | 0-3 Months, will be collected at 3 month visit
  Stereo Fly test
Stereoacuity | 3-6 Months, will be collected at 6 month visit
  Stereo Fly test
Ocular alignment | Baseline, will be collected at enrollment visit
  Alternative prism cover test at distance and at near
Ocular alignment | 0-3 Months, will be collected at 3 month visit
  Alternative prism cover test at distance and at near
Ocular alignment | 3-6 Months, will be collected at 6 month visit
  Alternative prism cover test at distance and at near
Near point of convergence | Baseline, will be collected at enrollment visit
  Near point of convergence (break point and recovery) will be measured using an accommodative target
Near point of convergence | 0-3 Months, will be collected at 3 month visit
  Near point of convergence (break point and recovery) will be measured using an accommodative target
Near point of convergence | 3-6 Months, will be collected at 6 month visit
  Near point of convergence (break point and recovery) will be measured using an accommodative target
Near visual acuity | Baseline, will be collected at enrollment visit
  Near visual acuity will be measured at 40 cm using the Rosenbaum card
Near visual acuity | 0-3 Months, will be collected at 3 month visit
  Near visual acuity will be measured at 40 cm using the Rosenbaum card
Near visual acuity | 3-6 Months, will be collected at 6 month visit
  Near visual acuity will be measured at 40 cm using the Rosenbaum card
Quality of Life Questionnaire- PedEyeQ | 0-3 Months, will be collected at 3 month visit
  Quality of life measures using the PedEyeQ
Quality of Life Questionnaire- PedEyeQ | 3-6 Months, will be collected at 6 month visit
  Quality of life measures using the PedEyeQ

IPD SHARING:
Plan to Share IPD: No